CLINICAL TRIAL: NCT05422989
Title: Public Health Risks and Characteristics of Upper Extremity Trauma During COVID-19 in the Gaza Strip: A Prospective Observational Study
Brief Title: Public Health Risks and Characteristics of Upper Extremity Trauma During COVID-19
Status: Completed | Type: Observational
Sponsor: Islamic University of Caza, Gaza, Palestine (Other)
Responsible Party: Principal Investigator, Najlaa M Abu Jamie, M.D, Islamic University of Caza, Gaza, Palestine
Other Study IDs: Upper Extremity Trauma
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Upper Extremity Injury; COVID-19
Keywords: Upper Extremity Trauma
MeSH Terms: conditions — Arm Injuries; COVID-19 | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: X-ray, CT — Just a diagnostic procedure to confirm the diagnosis

SUMMARY:
The aim of this study was to evaluate for the first time in the Gaza-strip the characteristics and incidence of Upper Extremity Trauma (UET) during the COVID-19 pandemic. The participants, investigated the characteristics of UET cases, and evaluated the UET primary medical-care. Additionally, also evaluate the obstacles in treating UET in Gaza during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Upper extremity trauma (UET) presenting to emergency departments (ED) incidence is rising. UET account for 20% to 40% of ED cases. UET affect daily function due to limited functionality of upper limb joints, nerves and muscles. The disability caused, affects psychological and social well-being, and major trauma may result in life changing long-term disability; Surgical site infection in UET is a possible cause of increased morbidity and mortality, leading to increased length of stay causing clinical and economic burden. UET in low income countries during armed conflict often causes a devastating decline in quality of life.

In the United States (U.S.), UET was estimated to be about 10% of all traumas, with 37.2 million cases, and estimated annual costs of 92 billion dollars; Over 2.7 million hand and wrist-related injuries/infections were presented to the ED nationwide; Pediatric nonballistic firearm UET cases in the U.S. represent a significant burden of disease. Electric scooters have also become an increasingly cause for UET. Interestingly, the current literature reflects a growing interest in sport related UET, as such sport related injuries may contribute to the growing incidence of UET worldwide.

The overall UET incidence among U.S. military personnel (n=214,993) was 15 per 1,000 person years (<1%); UET are a common cause of morbidity and disability affecting military readiness, and imposing an economic burden. According to the United Nations Office for the Coordination of Humanitarian Affairs 2019 report, 87% of about 7,500 injuries during 17 months were classified as UET; The report estimated that about 18.5% of the injured require specialized limb reconstruction treatment, with individual treatment costs up to US$ 40,000; Leaving the healthcare needs with a growing funding gap due to the high toll of UET.

UET reported during COVID-19 in the U.S. were significantly fewer in 2020 than in previous years; However, the odds of being admitted to the hospital when presenting with an UET were significantly greater. While traumatic injuries were less common during lockdowns, but the incidence of UET increased during COVID-19 quarantine in Italy. UET during COVID-19 quarantine was a predominantly male-disorder (over 60%)mostly due to domestic traumas.During other times, the affected population was younger and the most common mechanisms were sport and traffic-related injuries.

At the end of COVID-19 lockdowns a spike of UET incidence (158%) was reported in the United Kingdom due to young malesporting injuries predoninantly; Falls from <1.5 meters were the most common cause requiring surgical intervention. Additionally, UET operative volume increased during lockdowns in specialized trauma centers; and five types of behavior were identified as causes leading to those injuries that included (1) high-risk behavior and lawlessness, (2) virus-related suicidality , (3) lack of support due to social-distancing, (4) domestic renovations and carpentry, and (5) avoidance of health care facilities and delay in getting and treatment.

UET has a full spectrum of presentations ranging from simple lacerations and cellulitis to complex amputations and necrotizing infections As UET prevalence rises there is a need to develop evidence-based changes to facilitate better UET management. Currently there is no ideal classification for UET, and even less information is available regarding complex traumatic UET. A major dilemma is presented by UET that requiring choosing between limb salvage and amputation. Comorbidities, pre-injury function and social situation must be considered, as well as surgical considerations (as amputations may present more favorable functional and psychological prognosis compared to lengthy complex salvage surgeries with high risk of unfavorable complications). A viewpoint published in the midst of the COVID-19 pandemic stated that the public health infrastructural inadequacies led to a crisis in the Gaza-strip regarding sanitation, hygiene, waste treatment and water supply; Thus exposing Gaza's population to more epidemiological risks and disease outbreaks.

ELIGIBILITY:
Inclusion Criteria:

1. UET ED/ surgical ward admission;
2. Signed informed consent form to participate in this study.

Exclusion Criteria:

* Inability to consent or refusal to participate.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Upper Extremity trauma who arrived to ED and need addmission to the surgical ward
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Upper Extremity Trauma in the Gaza-Strip | Nine months
  Analysis of the public health Characteristics of UET during COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Yassin, M.D, Study Chair — Rabin Medical Center, Tel Aviv University School of Medicine, Israel.
Locations (1):
- Islamic University of Gaza, Gaza, Palestine, Israel

IPD SHARING:
Plan to Share IPD: No